CLINICAL TRIAL: NCT00000147
Title: Longitudinal Optic Neuritis Study (LONS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Masking: Single | Purpose: Treatment
Other Study IDs: NEI-48
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 1999-10

CONDITIONS: Multiple Sclerosis; Optic Neuritis
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis | interventions — Methylprednisolone; Prednisone

INTERVENTIONS:
Drug: Methylprednisolone
Drug: Prednisone

SUMMARY:
To assess the beneficial and adverse effects of corticosteroid treatment for optic neuritis.

To determine the natural history of vision in patients who suffer optic neuritis.

To identify risk factors for the development of multiple sclerosis in patients with optic neuritis.

DETAILED DESCRIPTION:
Optic neuritis is an inflammatory disease of the optic nerve that typically affects young adults. Women are affected more often than men. It is second only to glaucoma as the most common acquired optic nerve disorder in persons younger than age 50.

In this disorder, closely linked to multiple sclerosis, prognosis for visual recovery is generally good. However, return of visual function is almost never complete. After resolution of optic neuritis, virtually all patients show some signs of optic nerve damage, and most are symptomatic. Even when a patient's acuity recovers to 20/20, abnormalities frequently remain in other measures such as contrast sensitivity, color vision, and visual field.

Prior to the Optic Neuritis Treatment Trial (ONTT), well-established guidelines for treating optic neuritis did not exist. Although corticosteroids had been used to treat this disease, studies to demonstrate their effectiveness had not been satisfactory. Some experts advocated treatment with oral prednisone while others recommended no treatment. Anecdotal reports suggested that high-dose intravenous corticosteroids might be effective.

The association between optic neuritis and multiple sclerosis is well established. Optic neuritis may be the first manifestation of multiple sclerosis, or it may occur later in its course. A strong case can be made for "isolated" optic neuritis being a forme fruste of multiple sclerosis, based on similarities between the two in such epidemiologic factors as gender, age, geographic distributions, cerebrospinal fluid changes, histocompatibility data, magnetic resonance imaging (MRI) changes, and family history. The magnitude of the risk of multiple sclerosis after optic neuritis is uncertain. Previous studies have reported very disparate results, with the risk being reported to be as low as 13 percent and as high as 88 percent. The importance of risk factors such as age, gender, and MRI changes in predicting which patients with optic neuritis are most likely to develop multiple sclerosis also is unclear.

The treatment phase of the study was called the Optic Neuritis Treatment Trial (ONTT), whereas the current long-term followup phase is called the Longitudinal Optic Neuritis Study (LONS). The study is being conducted at 15 clinical centers in the United States. Resource centers include a data coordinating center and a visual field reading center.

Patients were randomized to one of the three following treatment groups at 15 clinical centers:

* Oral prednisone (1 mg/kg/day) for 14 days
* Intravenous methylprednisolone (250 mg every 6 hours) for 3 days, followed by oral prednisone (1 mg/kg/day) for 11 days
* Oral placebo for 14 days.

Each regimen was followed by a short oral taper. The oral prednisone and placebo groups were double masked, whereas the intravenous methylprednisolone group was single masked.

Baseline testing included blood tests to evaluate for syphilis and systemic lupus erythematosus, a chest x-ray to evaluate for sarcoidosis, and a brain MRI scan to evaluate for changes suggestive of multiple sclerosis.

The rate of visual recovery and the long-term visual outcome were both assessed by measures of visual acuity, contrast sensitivity, color vision, and visual field at baseline, at seven followup visits during the first 6 months, and then yearly. A standardized neurologic examination with an assessment of multiple sclerosis status was made at baseline, after 6 months, and then yearly.

ELIGIBILITY:
The major eligibility criteria for enrollment into the ONTT included the following:

Age range of 18 to 46 years

Acute unilateral optic neuritis with visual symptoms for 8 days or less

A relative afferent pupillary defect and a visual field defect in the affected eye

No previous episodes of optic neuritis in the affected eye

No previous corticosteroid treatment for optic neuritis or multiple sclerosis

No systemic disease other than multiple sclerosis that might be the cause of the optic neuritis

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1988-07

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of Arkansas, Little Rock, Arkansas
  - California Pacific Medical Center, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Illinois, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - New York University, New York, New York
  - Duke University, Durham, North Carolina
  - Devers Eye Institute, Portland, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Background] Beck RW; Diehl L; Cleary PA; Optic Neuritis Study Group; The Pelli-Robson Letter Chart: Normative data for young adults., Clin Vis Sci 1993;8:207-210
- [Background] Cleary PA, Beck RW, Anderson MM Jr, Kenny DJ, Backlund JY, Gilbert PR. Design, methods, and conduct of the Optic Neuritis Treatment Trial. Control Clin Trials. 1993 Apr;14(2):123-42. doi: 10.1016/0197-2456(93)90015-6. PMID 8500302
- [Background] Keltner JL, Johnson CA, Beck RW, Cleary PA, Spurr JO. Quality control functions of the Visual Field Reading Center (VFRC) for the Optic Neuritis Treatment Trial (ONTT). Control Clin Trials. 1993 Apr;14(2):143-59. doi: 10.1016/0197-2456(93)90016-7. PMID 8500303
- [Background] Anderson MM Jr, Boly LD, Beck RW. Remote clinic/patient monitoring for multicenter trials. Optic Neuritis Study Group. Control Clin Trials. 1996 Oct;17(5):407-14. doi: 10.1016/s0197-2456(96)00021-9. PMID 8932973
- [Background] Optic Neuritis Study Group; The five-year risk of multiple sclerosis after optic neuritis. Experience of the Optic Neuritis Treatment Trial., Neurology (in press)
- [Background] Visual function 5 years after optic neuritis: experience of the Optic Neuritis Treatment Trial. The Optic Neuritis Study Group. Arch Ophthalmol. 1997 Dec;115(12):1545-52. PMID 9400788
- [Background] The clinical profile of optic neuritis. Experience of the Optic Neuritis Treatment Trial. Optic Neuritis Study Group. Arch Ophthalmol. 1991 Dec;109(12):1673-8. doi: 10.1001/archopht.1991.01080120057025. PMID 1841573
- [Background] Beck RW, Cleary PA, Anderson MM Jr, Keltner JL, Shults WT, Kaufman DI, Buckley EG, Corbett JJ, Kupersmith MJ, Miller NR, et al. A randomized, controlled trial of corticosteroids in the treatment of acute optic neuritis. The Optic Neuritis Study Group. N Engl J Med. 1992 Feb 27;326(9):581-8. doi: 10.1056/NEJM199202273260901. PMID 1734247
- [Background] Beck RW. Corticosteroid treatment of optic neuritis: a need to change treatment practices. The Optic Neuritis Study Group. Neurology. 1992 Jun;42(6):1133-5. doi: 10.1212/wnl.42.6.1133. No abstract available. PMID 1318520
- [Background] Beck RW. The optic neuritis treatment trial. Implications for clinical practice. Optic Neuritis Study Group. Arch Ophthalmol. 1992 Mar;110(3):331-2. doi: 10.1001/archopht.1992.01080150029020. No abstract available. PMID 1543448
- [Background] Beck RW, Arrington J, Murtagh FR, Cleary PA, Kaufman DI. Brain magnetic resonance imaging in acute optic neuritis. Experience of the Optic Neuritis Study Group. Arch Neurol. 1993 Aug;50(8):841-6. doi: 10.1001/archneur.1993.00540080050013. PMID 8352671
- [Background] Beck RW, Cleary PA. Optic neuritis treatment trial. One-year follow-up results. Arch Ophthalmol. 1993 Jun;111(6):773-5. doi: 10.1001/archopht.1993.01090060061023. PMID 8512477
- [Background] Beck RW, Cleary PA. Recovery from severe visual loss in optic neuritis. Arch Ophthalmol. 1993 Mar;111(3):300. doi: 10.1001/archopht.1993.01090030018009. No abstract available. PMID 8447730
- [Background] Beck RW, Cleary PA, Trobe JD, Kaufman DI, Kupersmith MJ, Paty DW, Brown CH. The effect of corticosteroids for acute optic neuritis on the subsequent development of multiple sclerosis. The Optic Neuritis Study Group. N Engl J Med. 1993 Dec 9;329(24):1764-9. doi: 10.1056/NEJM199312093292403. PMID 8232485
- [Background] Beck RW, Kupersmith MJ, Cleary PA, Katz B. Fellow eye abnormalities in acute unilateral optic neuritis. Experience of the optic neuritis treatment trial. Ophthalmology. 1993 May;100(5):691-7; discussion 697-8. doi: 10.1016/s0161-6420(13)31589-9. PMID 8493012
- [Background] Chrousos GA, Kattah JC, Beck RW, Cleary PA. Side effects of glucocorticoid treatment. Experience of the Optic Neuritis Treatment Trial. JAMA. 1993 Apr 28;269(16):2110-2. PMID 8468765
- [Background] Keltner JL, Johnson CA, Spurr JO, Beck RW. Baseline visual field profile of optic neuritis. The experience of the optic neuritis treatment trial. Optic Neuritis Study Group. Arch Ophthalmol. 1993 Feb;111(2):231-4. doi: 10.1001/archopht.1993.01090020085029. PMID 8431161
- [Background] Beck RW, Cleary PA, Backlund JC. The course of visual recovery after optic neuritis. Experience of the Optic Neuritis Treatment Trial. Ophthalmology. 1994 Nov;101(11):1771-8. doi: 10.1016/s0161-6420(94)31103-1. PMID 7800355
- [Background] Keltner JL, Johnson CA, Spurr JO, Beck RW. Visual field profile of optic neuritis. One-year follow-up in the Optic Neuritis Treatment Trial. Arch Ophthalmol. 1994 Jul;112(7):946-53. doi: 10.1001/archopht.1994.01090190094027. PMID 8031275
- [Background] Beck RW. The optic neuritis treatment trial: three-year follow-up results. Arch Ophthalmol. 1995 Feb;113(2):136-7. doi: 10.1001/archopht.1995.01100020014004. No abstract available. PMID 7864737
- [Background] Beck RW, Trobe JD. The Optic Neuritis Treatment Trial. Putting the results in perspective. The Optic Neuritis Study Group. J Neuroophthalmol. 1995 Sep;15(3):131-5. No abstract available. PMID 8574355
- [Background] Beck RW, Trobe JD. What we have learned from the Optic Neuritis Treatment Trial. Ophthalmology. 1995 Oct;102(10):1504-8. doi: 10.1016/s0161-6420(95)30839-1. No abstract available. PMID 9097798
- [Background] Rolak LA, Beck RW, Paty DW, Tourtellotte WW, Whitaker JN, Rudick RA. Cerebrospinal fluid in acute optic neuritis: experience of the optic neuritis treatment trial. Neurology. 1996 Feb;46(2):368-72. doi: 10.1212/wnl.46.2.368. PMID 8614496
- [Background] Trobe JD, Beck RW, Moke PS, Cleary PA. Contrast sensitivity and other vision tests in the optic neuritis treatment trial. Am J Ophthalmol. 1996 May;121(5):547-53. doi: 10.1016/s0002-9394(14)75429-7. PMID 8610798
- [Background] Cleary PA, Beck RW, Bourque LB, Backlund JC, Miskala PH. Visual symptoms after optic neuritis. Results from the Optic Neuritis Treatment Trial. J Neuroophthalmol. 1997 Mar;17(1):18-23; quiz 24-8. doi: 10.1016/s0002-9394(14)70814-1. PMID 9093956